CLINICAL TRIAL: NCT00904345
Title: Phase II Study of RT Concurrent w/ Cetuximab in Patients w/ Locally Advanced Head & Neck SCC Who Do Not Qualify For Standard Chemotherapy Due To Age >70 Or Co-Morbidities
Brief Title: Study of Radiation (RT) Concurrent With Cetuximab in Patients With Advanced Head and Neck Squamous Cell Carcinoma (SCC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopped early for funding and efficacy reasons.
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2009.009; HUM 27253 (Other: University of Michigan Medical IRB); NCT01250522 (obsolete NCT alias)
Record Dates: First submitted 2009-05-17; First posted 2009-05-19 (Estimated); Results first posted 2021-01-20 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Head and Neck Cancer
Keywords: SCC Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Cetuximab; Radiation: 50-60 Gy and 70 Gy

INTERVENTIONS:
Drug: Cetuximab — Patients will receive a single dose of cetuximab 400 mg/m (Day 0). On day 7 (+/- 1 day), a repeat biopsy will be performed. Radiation concurrent with weekly cetuximab 250 mg/m.
Radiation: 50-60 Gy and 70 Gy — Within approximately 4 days (after single dose of Cetuximab), definitive radiation will begin (70 Gy in 35 fractions to the gross tumor, 50-60 Gy to subclinical target volumes) concurrent with weekly cetuximab 250 mg/m.

SUMMARY:
This is a single-arm, phase II trial to characterize the clinical outcome of standard of care, cetuximab concurrent with radiation, in a special population (head and neck cancer patients who cannot tolerate concurrent chemoradiotherapy due to advanced age, poor performance status or concurrent illness), and to determine if biomarker response to a loading dose of cetuximab is predictive of that outcome.

DETAILED DESCRIPTION:
Primary Objective 1: Determine changes in tumor EGFR, pEGFR, downstream signaling and novel phosphoproteins following a loading dose of cetuximab in patients who are poor candidates for chemoradiation (age =70 years or with significant co-morbidities) and are therefore treated with cetuximab with radiation.

Primary Objective 2: Characterize clinical outcomes, including local recurrence, progression-free survival and overall survival in these patients, and correlate these clinical outcomes with the changes in tumor EGFR, pEGFR, downstream signaling, and novel phosphoproteins.

Primary Objective 3: Describe the toxicity, in particular mucositis/dysphagia, of this regimen.

Secondary Objective 1: Conduct normal mucosa EGFR assessment for comparison with tumor sample.

Secondary Objective 2: Correlate HPV presence and titer with p53 status and clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically-confirmed, previously untreated, clinically accessible (without general anesthesia) locally advanced squamous cell carcinoma of the larynx, hypopharynx, oropharynx, oral cavity, or nonresectable head and neck squamous cell carcinomas of the skin.
* Patients will be limited to:

  * ≥ 70 years of age, OR
  * with co-morbidities that preclude treatment with standard platinum-based chemotherapy, as determined by the treating physician, OR
  * KPS ≤ 80, OR
  * Creatinine clearance < 30 cc/min
* Laboratory criteria:

  * WBC > 3500/ul
  * Granulocyte > 1500/ul
  * Platelet count > 100,000/ul
  * Total Bilirubin < 1.5 X ULN
  * AST and ALT < 2.5 X ULN
* Patients must give documented informed consent to participate in this study.

Exclusion Criteria:

* Prior head and neck malignancy, or history of other prior non-head and neck malignancy within the past 3 years (excluding skin cancer and early stage treated prostate cancer).
* Prior head and neck radiation or chemotherapy.
* Documented evidence of distant metastases.
* Patients with nasopharyngeal carcinoma.
* Any medical or psychiatric illness, which, in the opinion of the principal investigator, would compromise the patient's ability to tolerate this treatment.
* Patients with psychiatric/social situations that would limit compliance with study requirements are not eligible.
* Patients with prior anti-epidermal growth-factor receptor antibody therapy (antibody or small molecule).
* Patients residing in prison.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-04; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shruti Jolly, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (2):
- United States (2):
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Michigan Veterans Administration Hospital, Ann Arbor, Michigan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 participants withdrew before receiving treatment
Groups:
- Treatment With Cetuximab + RT: Patients received a single loading dose of cetuximab 400 mg/m (Day 0), then weekly cetuximab 250 mg/m concurrent with radiation. Within approximately 4 days after first (loading) dose of cetuximab, patients received radiation administered as 70 Gy in 35 fractions to the gross tumor, 50-60 Gy to subclinical target volumes.
Period: Overall Study
Arm/Group | Treatment With Cetuximab + RT
Started | 21
Stopped or Modified Treatment Due to Toxicity | 3
Completed (18 completed treatment with RT + Cetuximab) | 18
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Treatment: Cetuximab + RT: Patients received a single loading dose of cetuximab and a cetuximab infusion delivered once a week during radiotherapy.
Arm/Group | Treatment: Cetuximab + RT
Number analyzed (Participants) | 21
Age, Continuous [Mean (Full Range); unit: years] | 65.6 [39 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 6
Smoking Status [Count of Participants; unit: Participants]
  Yes, current | 7
  Yes, past | 13
  No | 1
Cancer Location [Count of Participants; unit: Participants]
  Oropharynx | 16
  Oral Cavity | 2
  Auditory Canal | 1
  Hypopharynx | 1
  Unknown primary | 1
HPV Status [Count of Participants; unit: Participants]
  Positive | 10
  Negative | 6
  Unknown | 5

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Tumor Epidermal Growth Factor Receptor (EGFR)
Description: The ratio (fold change) of tumor EGFR post-loading dose/pre-loading dose of cetuximab. Reported as the mean of fold changes across all participants who had an evaluable tumor sample.
Time Frame: At baseline (pre-loading dose) and day 7 post-loading dose
Population: 15 participants had a sample size sufficient for EGFR analysis.
Measure: Mean (Full Range); unit: fold change
Arm/Group | Treatment: Cetuximab + RT
Number analyzed (Participants) | 15
fold change | 0.56 [0 to 1.1]

2. Primary Outcome: Mean Change in Tumor Phosphorylated EGFR (pEGFR)
Description: The ratio (fold change) of tumor pEGFR post-loading dose/pre-loading dose of cetuximab. Reported as the mean of fold changes across all participants who had an evaluable tumor sample.
Time Frame: At baseline (pre-loading dose) and day 7 post-loading dose
Population: 10 participants had a sample size sufficient for pEGFR analysis.
Measure: Mean (Full Range); unit: fold change
Arm/Group | Treatment: Cetuximab + RT
Number analyzed (Participants) | 10
fold change | 0.81 [0 to 3]

3. Primary Outcome: Progression Free Survival Rate
Description: Percentage of participants who survived without recurrent disease, from the time of enrollment to 1 and 2 years.
Time Frame: At 1 and 2 years
Population: Patients who completed the full course of cetuximab+RT or had cetuximab+RT stopped for toxicity.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment: Cetuximab + RT
Number analyzed (Participants) | 21
percentage of participants
  1 year | 47.8 [29.9 to 76.5]
  2 year | 37.2 [20.7 to 66.8]
Statistical Analysis 1: Comparison: Treatment: Cetuximab + RT; Test type: Other; Estimates of proportion event-free at 1 and 2 years calculated using Kaplan-Meier methods, and the 2-sided, 95% confidence intervals were calculated by the Greenwood method. All analyses were performed using SAS v9.4 software and R version 3.5.2

4. Primary Outcome: Overall Survival Rate
Description: Percentage of participants alive at 1 and 2 years after enrollment.
Time Frame: At 1 and 2 Years
Population: Patients who completed the full course of cetuximab+RT or had cetuximab+RT stopped for toxicity.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment: Cetuximab + RT
Number analyzed (Participants) | 21
percentage of participants
  1 year | 68.8 [50.9 to 93]
  2 years | 47.6 [29.7 to 76.3]
Statistical Analysis 1: Comparison: Treatment: Cetuximab + RT; Test type: Other; Survival proportion estimates at 1 and 2 years were calculated using Kaplan-Meier methods, and the 2-sided, 95% confidence intervals calculated by the Greenwood method. All analyses were performed using SAS v9.4 software and R version 3.5.2

5. Primary Outcome: Number of Participants With Treatment Related Toxicities
Description: Toxicities are measured by number of participants who experience one or more types or indicator of toxicity, shown as all grades and grades 3-4. As each participant could have multiple toxicities, the total number of incidents outnumbers the number of participants. Toxicities are graded according to the CTCAE v4.
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Treatment: Cetuximab + RT
Number analyzed (Participants) | 21
participants
  All Grades: Cutaneous Toxicity | 16
  All Grades: Mucositis | 19
  All grades: Dysphagia | 14
  All grades: Hematologic Toxicity | 3
  Grades 3-4: Cutaneous Toxicity | 4
  Grades 3-4: Mucositis | 8
  Grades 3-4: Dysphagia | 5
  Grades 3-4: Hematologic Toxicity | 0

6. Secondary Outcome: Change in Tumor EGFR Level Relative to EGFR in Normal Mucosa
Description: Normal mucosa EGFR was assessed for comparison with EGFR in tumor sample. The fold change in tumor EGFR level at post-loading dose/pre-loading dose of cetuximab, relative to fold change in normal mucosa EGFR level post-loading dose/pre-loading dose of cetuximab was summarized across all participants who had an evaluable tumor sample and normal mucosa sample. The value reported is the ratio of fold change in tumor/fold change in buccal EGFR.
Time Frame: At baseline (pre-loading dose) and day 7 post-loading dose
Population: 6 participants had a sample size sufficient for EGFR analysis.
Measure: Mean (Full Range); unit: ratio
Arm/Group | Treatment: Cetuximab + RT
Number analyzed (Participants) | 6
ratio | 0.84 [0 to 2.2]

7. Secondary Outcome: Change in Tumor pEGFR Level Relative to pEGFR in Normal Mucosa
Description: Normal mucosa pEGFR was assessed for comparison with pEGFR in tumor sample. The fold change in tumor pEGFR level post-loading dose/pre loading dose of cetuximab, relative to fold change in normal mucosa pEGFR level post-loading dose/pre-loading dose of cetuximab was summarized across all participants who had an evaluable tumor sample and normal mucosa sample. The value reported is the ratio of fold change in tumor/fold change in buccal pEGFR.
Time Frame: At baseline (pre-loading dose) and day 7 post-loading dose
Population: 7 participants had a sample size sufficient for pEGFR analysis.
Measure: Mean (Full Range); unit: ratio
Arm/Group | Treatment: Cetuximab + RT
Number analyzed (Participants) | 7
ratio | 4.69 [0 to 30]

8. Post Hoc Outcome: Freedom From Local Regional Progression (FFLRP)
Description: Percentage of participants without local or regional failure from the time of enrollment to 1 and 2 years.
Time Frame: At 1 and 2 years
Population: Patients who completed the full course of cetuximab+RT or had cetuximab+RT stopped for toxicity.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment: Cetuximab + RT
Number analyzed (Participants) | 21
percentage of participants
  1 year | 63.9 [44.5 to 92]
  2 years | 51.2 [31.7 to 82.5]
Statistical Analysis 1: Comparison: Treatment: Cetuximab + RT; Test type: Other; Estimates of proportion LRP event-free at 1 and 2 years were calculated using Kaplan-Meier methods, and the 2-sided, 95% confidence intervals calculated by the Greenwood method. All analyses were performed using SAS v9.4 software and R version 3.5.2

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Treatment: Cetuximab + RT
All-Cause Mortality (participants affected / at risk) | 12/21
Serious Adverse Events (participants affected / at risk) | 12/21
Other Adverse Events (participants affected / at risk) | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment: Cetuximab + RT (N=21)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 3 (4)
Esophagitis (Gastrointestinal disorders) | 1 (2)
Gastrointestinal disorders - Unspecified (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (4)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 2 (2)
Skin infection (Infections and infestations) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Delirium (Psychiatric disorders) | 1 (1)
Psychiatric disorders - Unspecified (Psychiatric disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment: Cetuximab + RT (N=21)
Anemia (Blood and lymphatic system disorders) | 3 (6)
Blood and lymphatic system disorders - Unspecified (Blood and lymphatic system disorders) | 2 (5)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 19 (50)
Dysphagia (Gastrointestinal disorders) | 16 (49)
Esophagitis (Gastrointestinal disorders) | 16 (24)
Gastrointestinal disorders - Unspecified (Gastrointestinal disorders) | 3 (6)
Mucositis oral (Gastrointestinal disorders) | 20 (52)
Nausea (Gastrointestinal disorders) | 7 (9)
Oral pain (Gastrointestinal disorders) | 4 (5)
Salivary duct inflammation (Gastrointestinal disorders) | 9 (33)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Chills (General disorders) | 2 (2)
Fatigue (General disorders) | 7 (7)
Fever (General disorders) | 2 (2)
Pain (General disorders) | 2 (3)
Papulopustular rash (Infections and infestations) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 17 (35)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (4)
Creatinine increased (Investigations) | 1 (2)
Lymphocyte count decreased (Investigations) | 3 (6)
Platelet count decreased (Investigations) | 1 (4)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 10 (17)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 6 (11)
Dysgeusia (Nervous system disorders) | 19 (48)
Facial muscle weakness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Myelitis (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Psychiatric disorders - Unspecified (Psychiatric disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (15)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 10 (16)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Unspecified (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/45/NCT00904345/Prot_SAP_000.pdf